CLINICAL TRIAL: NCT05837429
Title: Comparison of the Effects of Continuous Aerobic Exercise Training and Low Volume High Intensity Interval Training on Cardiopulmonary Exercise Capacity, Autonomic Function and Oxidative Stress in Operated Lung Cancer Patients
Brief Title: Low Volume High Intensity Interval Training in Operated Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Hamide Sahin-Yildiz, Principal Investigator, PT, Msc, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-194-22
Record Dates: First submitted 2023-04-15; First posted 2023-05-01 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: Low volume high intensity interval training; Aerobic exercise; Oxidative stress; Cardiopulmonary exercise test
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Volume High Intensity Exercise Training (Experimental): Patients in the intervention group will be given a warm-up phase for 3 minutes at 50% VO2max, 1 minute at 80-100% VO2max and 1 minute at 50% VO2max in 10 cycles, and finally a cool-down phase for 3 minutes at 50% VO2max.
  Interventions: Behavioral: Low Volume High Intensity Exercise Training
- Aerobic Exercise (Active Comparator): Patients in the control group will be given exercise training on a bicycle ergometer for 5 minutes warm-up phase at 40% of maximal oxygen consumption (VO2max), 20 minutes exercise phase at 60% of VO2max and 5 minutes cool down phase at 40% of VO2max for a total of 30 minutes.
  Interventions: Behavioral: Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Low Volume High Intensity Exercise Training — Patients in the intervention group will be given a warm-up phase for 3 minutes at 50% VO2max, 1 minute at 80-100% VO2max and 1 minute at 50% VO2max in 10 cycles, and finally a cool-down phase for 3 minutes at 50% VO2max.
  Arms: Low Volume High Intensity Exercise Training
Behavioral: Aerobic Exercise Training — Patients in the control group will be given exercise training on a bicycle ergometer for 5 minutes warm-up phase at 40% of maximal oxygen consumption (VO2max), 20 minutes exercise phase at 60% of VO2max and 5 minutes cool down phase at 40% of VO2max for a total of 30 minutes.
  Arms: Aerobic Exercise

SUMMARY:
Patients included in the study will be randomly divided into 2 groups using appropriate randomization programs. All patients will be given exercise training individually for 24 sessions using a bicycle ergometer under the supervision of a physiotherapist.Patients in the first group will be given exercise training on a bicycle ergometer for 5 minutes warm-up phase at 40% of maximal oxygen consumption (VO2max), 20 minutes exercise phase at 60% of VO2max and 5 minutes cool down phase at 40% of VO2max for a total of 30 minutes. Patients in the second group will be given a warm-up phase for 3 minutes at 50% VO2max, 1 minute at 80-100% VO2max and 1 minute at 50% VO2max in 10 cycles, and finally a cool-down phase for 3 minutes at 50% VO2max. In total, 25 minutes of low-volume high-intensity intermittent exercise training will be given on a bicycle ergometer.

DETAILED DESCRIPTION:
The study will include patients diagnosed with non-small cell lung cancer who have completed adjuvant treatments such as chemotherapy and radiotherapy at least 6 months ago, stage 3A or earlier,clinically stable remission (no recurrence or active cancer), and have been followed by Ankara University Medical Oncology Department. Patients who have undergone pneumonectomy surgery, patients with advanced COPD and cardiac disease, patients with orthopedic or neurological problems who cannot adapt to exercise will be excluded. Patients included in the study will be randomly divided into 2 groups using appropriate randomization programs. All patients will be given exercise training individually for 24 sessions using a bicycle ergometer under the supervision of a physiotherapist. To determine the intensity of exercise training, all patients will undergo Cardiopulmonary Exercise Test (CPET) on a bicycle ergometer under the supervision of a physiotherapist and a physician before the training sessions. During CPET, maximal oxygen capacity, diffusion capacity, heart rate variability as a marker of autonomic function and heart rate recovery will be measured. Patients in the first group will be given exercise training on a bicycle ergometer for 5 minutes warm-up phase at 40% of maximal oxygen consumption (VO2max), 20 minutes exercise phase at 60% of VO2max and 5 minutes cool down phase at 40% of VO2max for a total of 30 minutes. Patients in the second group will be given a warm-up phase for 3 minutes at 50% VO2max, 1 minute at 80-100% VO2max and 1 minute at 50% VO2max in 10 cycles, and finally a cool-down phase for 3 minutes at 50% VO2max. In total, 25 minutes of low-volume high-intensity intermittent exercise training will be given on a bicycle ergometer. After the exercise training, CPET will be performed again in the presence of a physician and physiotherapist to evaluate the effectiveness of the exercise. Blood samples of all groups will be taken by the physician before and after training to obtain information about the change in oxidative stress (total oxidant status, total antioxidant status) and myokine (irisin hormone) biomarkers between the two exercise modalities. Knee extensors and hand grip strength will be evaluated with a dynamometer as part of the peripheral muscle strength assessment of all groups before and after the training. EORTC QLQ-C30 quality of life questionnaire and London Chest Activities of Daily Living Scale will be used to evaluate the effect of exercise training on quality of life and activities of daily living before and after training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Non-Small Cell Lung Cancer
* Stage 3A and earlier
* Operated and at least 6 months have expired since the surgery
* Having completed adjuvant treatments such as chemotherapy and radiotherapy and at least 6 months have expired
* Being clinically stable and in remission
* Not having new recurrence and active cancer

Exclusion Criteria:

* Pneumonectomy surgery
* Presence of symptoms, signs and diagnoses indicating the presence of lung and cardiac disease such as advanced COPD
* Having any orthopedic or neurological problem that may prevent exercise
* Presence of recurrence or active cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-04-06 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption | 24 months
  To be measured during cardiopulmonary exercise testing
Heart Rate Variability | 24 months
  To be measured during cardiopulmonary exercise testing
Oxidative Stress | 24 months
  Lipid peroxidation marker from serum for determination of oxidative damage melondialdehyde (MDA), total oxidant status (TOS), total antioxidant status (TAS) parameters will be evaluated.
Myokine | 24 months
  Irisin levels in serum, enzyme-linked immunosorbent assay (Enzyme-Linked Immuno Sorbent Assay-ELISA) method using a commercial kit.

SECONDARY OUTCOMES:
Change in quality of life | 24 months
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire QLQ-C30 will be used for quality of life assessment. Higher scores reflect better function, whereas lower scores suggest impairment.
Peripheral Muscle Strength | 24 months
  The strength of the knee extensors will be measure using a digital dynamometer (Lafayette, Lafayette Instrument, Lafayette, IN, USA). The test will repeat 3 times on the dominant side and recorded in kilograms (kg). A Jamar hand dynamometer (Fabrication Enterprises, New York, USA) will be use to measure the handgrip strength. The measurement will repeat 3 times on the dominant side and recorded in kg.
Activity of Daily Living | 24 months
  London Chest Activity of Daily Living Scale will be used for activity of daily living assessment. Low scores represent high activity.

CONTACTS AND LOCATIONS:
Overall Officials: Hamide Sahin-Yildiz, Msc,PT, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No